CLINICAL TRIAL: NCT06276270
Title: Multi-centre, Open-label, First-in-man Study With Mucopad HA Used in Adult Patients Suffered From Oral Mucositis After Radiotherapy
Brief Title: Multi-centre, Open-label, First-in-man Study With Mucopad HA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Contipro Pharma a.s. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PT-MUC-1_05-21
Record Dates: First submitted 2024-02-14; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device is administered directly onto the area affected by mucositis. (Experimental)
  Interventions: Device: Mucopad HA

INTERVENTIONS:
Device: Mucopad HA — The product is a Class III Medical Device incorporating a medicinal substance (antiseptics-octenidine) within the composition made of sodium hyaluronate polysacharide stabilised by calcium chloride. Device is administered directly onto the area affected by mucositis.

SUMMARY:
The device´s intended use is to treat defects and/or lesions of the oral mucosa, e.g. oral mucositis.To prove safety of the device in terms of clinical results.

DETAILED DESCRIPTION:
This is an multi-centre, open-label, first-in-man prospective study.

Up to 60 patients in total will be involved in the open-label trial of new medical device - Mucopad HA. Eligible patients will be undergoing treatment with the device for up to 10 weeks, after which it is expected that there should be significant improvement in the healing process of oral mucositis after radiotherapy. It is considered as an improvement when there is a significant reduction or complete resolution of the mucositis. Mucositis will be assessed as a WHO scale.

Quality of life will be assessed by Oral Mucositis Daily Questionnaire (OMDQ) provided by FACIT. The FACIT and all related works are owned and copyrighted by, and the intellectual property of David Cella, Ph.D. Permission for use of the OMDQ questionnaire is obtained by contacting Dr. Cella at information@facit.org.

List of investigational sites is in appendix 7.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Oral Mucositis after radiotherapy of grade I - IV according to WHO
* Patient willing and able to provide the written consent
* Ability to communicate well with the investigator in the local language, and to understand and comply with the requirements of the study

Exclusion Criteria:

* Age < 18 years
* Pregnant or lactating women
* Patients in terminal stage of living
* Patients with known hypersensitivity or allergy to any of the substances contained in Medical Device
* Alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Resolution of mucositis symptoms since completion of radiotherapy | 10 weeks
  healing time

SECONDARY OUTCOMES:
- Pain management (VAS scale) | 10 weeks
  pain value 1-100
Development of xerostomy | 10 weeks
  xerostomy yes/no
Subjective evaluation on scale 1-5 of the treatment by investigator/ patient | 10 weeks
  scale 1-5

CONTACTS AND LOCATIONS:
Locations (5):
- Czechia (5):
  - Masarykův onkologický ústav, Klinika radiační onkologie, Brno, Česká Republika
  - FN Hradec Králové Klinika onkologie a radioterapie, Hradec Králové, Česká Republika
  - Fakultní nemocnice Ostrava, Klinika onkologická, Ostrava, Česká Republika
  - Etická komise FN Bulovka, Prague, Česká Republika
  - Fakultní Thomayerova nemocnice Onkologická klinika 1.LF UK a FTN, Prague, Česká Republika

IPD SHARING:
Plan to Share IPD: No